CLINICAL TRIAL: NCT05574114
Title: A Phase I Study Of Split-Course Bridging Radiotherapy (SC-BRT) Prior To Commercial CD19 CAR T-Cell Therapies For Patients With Relapsed or Refractory B-Cell Lymphomas
Brief Title: A Study of Radiation Therapy Before CAR T Cell Therapy for People With B Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 22-217
Record Dates: First submitted 2022-10-06; First posted 2022-10-10 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Non-Hodgkin Lymphoma; Non-Hodgkin's Lymphoma, Relapsed; Non-Hodgkin's Lymphoma Refractory
Keywords: Split-Course Bridging Radiotherapy; CD19 CAR T-Cell Therapies; 22-217
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Recurrence

STUDY DESIGN:
Intervention Model Description: This is a single arm, Phase I trial designed to describe the feasibility and safety of a standardized, stage-adapted, split-course BRT regimen prior to standard of care, commercial anti-CD19 CAR T-cell therapy. This design incorporates a small early safety cohort with the option for a potential patient expansion cohort.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radiation Therapy Before CAR T Cell Therapy (Experimental): For the purposes of this protocol, day 0 will be considered the date of planned CAR T infusion. BRT Part I (intervention is 9 fractions of 3 Gy to a total dose of 27 Gy). Post-BRT Phase I re- evaluation period: Following delivery of the first 9- fractions of BRT, patients will have a period for recovery, and undergo protocol-mandated reassessment (e.g., PET scan and biopsy). Patients will receive standard of care lymphodepleting chemotherapy. Substitutions to the lymphodepleting regimen will be permitted at the discretion of the treating investigator. Day -2: BRT Part II (intervention is one fraction 3 Gy to receive a total dose of 3 Gy). Day -1: No protocol scheduled treatment interventions. Day 0: Subject will receive standard of care infusion of a manufactured commercial CAR T-cell product, as an inpatient or outpatient, at the discretion of the treating investigator.
  Interventions: Radiation: Bridging radiotherapy (BRT); Drug: Conditioning chemotherapy; Biological: CAR T-cell product

INTERVENTIONS:
Radiation: Bridging radiotherapy (BRT) — RT Part I. The target will be to complete the 9th fraction of radiotherapy (i.e., total of 27Gy) between days -12 and -8 Day -2: BRT Part II (intervention is one fraction 3 Gy to receive a total dose of 3 Gy).
Drug: Conditioning chemotherapy — Day -5 to -3: Patients will receive standard of care lymphodepleting chemotherapy
Biological: CAR T-cell product — Day 0: Subject will receive standard of care infusion of a manufactured commercial CAR T-cell product.

SUMMARY:
The purpose of this study is to test whether radiation therapy given before standard CAR T cell therapy is a safe and effective treatment for people with relapsed and refractory B cell lymphoma. The researchers will also study whether radiation therapy used in this study is a practical treatment option before standard CAR T cell therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, relapsed or refractory non-Hodgkin lymphoma patients eligible for a CAR T-cell therapy, such as DLBCL (including transformed follicular lymphoma), high grade B-cell lymphoma, primary mediastinal B-cell lymphoma, and follicular lymphoma of any grade
* Patient is approved for, and planned to receive, anyone of the three commercially available anti-CD19 CAR T-cell products (axicabtagene ciloleucel, maraleucel or tisagenlecleucel)
* Patient has at least one site of disease with avidity greater than liver on a screening FDG-PET scan performed within 2 months of RT simulation. Measurable disease is not required.
* Active secondary central nervous system (CNS) lymphoma is allowed
* Age 18 or older
* ECOG status ≤2
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile or abstain from sexual activity for the course of the study through 120 days after the last dose of radiotherapy. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year. Note: Abstinence is acceptable if this is the established and preferred contraception for the subject
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy. Note: Abstinence is acceptable if this is the established and preferred contraception for the subject

Exclusion Criteria:

* Subject is planned to receive any systemic therapy after initiation of BRT and before re-infusion of CAR T cells including conventional chemotherapy, immunotherapy or targeted agents [Note: Planned lymphodepletion chemotherapy in preparation for CAR T cell administration is not an exclusion criterion]
* Subject has received prior RT to any site(s) planned for bridging therapy such that the composite dose considering the protocol-mandated BRT would exceed normal tissue tolerances in the determination of the investigator.
* The treating investigator deems that it would be impossible to comprehensively treat the patient with radiotherapy given concerns about feasibility or potential toxicities
* Current or planned pregnancy
* Known additional malignancy that is progressing or requires any treatment other than active surveillance or hormonal therapy. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Subject has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study based on the investigator´s judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
number of patients who develop unanticipated severe toxicity events | 1 year
  Reporting of toxicities will be based on Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 except for CRS and ICANS which will be evaluated using ASTCT Consensus grading.

SECONDARY OUTCOMES:
number of patients who are able to receive comprehensive BRT prior to infusion of CAR T cells | 2 years
  Comprehensive is defined as delivery of high- or low-dose RT to all sites of PET-avid disease.

CONTACTS AND LOCATIONS:
Overall Officials: Lia Palomba, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm